CLINICAL TRIAL: NCT05843721
Title: An Open Post-marketing Clinical Follow-up Investigation to Follow Long-term Performance and Safety of Intranasal Kinetic Oscillation in Subjects With Chronic Migraine
Brief Title: Post-marketing Clinical Follow-up for Long-term Use of Intranasal Kinetic Oscillation in Subjects With Chronic Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties recruiting patients in combination with good results in data analysis.
Sponsor: Chordate Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PM010
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KOS treatment (Other): Treatment with intranasal kinetic oscillation stimulation (KOS)
  Interventions: Device: KOS (Intranasal kinetic oscillation stimulation)

INTERVENTIONS:
Device: KOS (Intranasal kinetic oscillation stimulation) — Treatment is 10 minutes in each nasal cavity. Totally 2 x 10 minutes per treatment.

SUMMARY:
An non controlled, long term, multi center investigation

DETAILED DESCRIPTION:
Subjects who provided written informed consent and are eligible for the study will be asked to complete a daily diary for 4 weeks during the screening period. In the diary the subjects will record headache and migraine days, any changes in their health, and concomitant medications they may be using. The data collected in the diary during this screening period will be used as Baseline for the performance assessments.

A non-controlled, long term, multi-center investigation for symptom improvement in subjects suffering headache and migraine attacks.

During the run-in (baseline) period and through the whole study the subjects will continue using their existing prescribed or over the counter (OTC) treatments.

Following the run-in period (4 weeks) the subjects will be treated six times within a period that is approximately 6 weeks. The first treatment will be given the first day after the run-in period.

During 12-month follow-up period (from the time of the first treatment), subjects will be treated when needed but a maximum of 14 treatments.

ELIGIBILITY:
INCLUSION AND EXCLUSION CRITERIA:

Inclusion Criteria

1. The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the informed consent form;
2. Male or female aged between 18 and 70 years (inclusive) at the time of providing informed consent;
3. Diagnosed with chronic migraine with or without aura (≥15 headache days per month including at least 8 migraine days for more than 3 months before screening) according to the International Headache Society classification (International Classification of Headache Disorders III);
4. Migraine onset before the age of 65 years;
5. Reported history of migraine for at least 1 year before screening;
6. Able and willing to maintain current prophylactic migraine medication regimen (if any) (no change in type, frequency or dose) from screening to at least the 6-month follow-up;
7. Women of childbearing potential must be willing to use highly effective contraceptive methods (failure rate <1% per year when used consistently and correctly) during the study.

Exclusion Criteria

1. Unable to distinguish between migraine headache and other headache types;
2. An ongoing upper respiratory infection, nasal tumors, or wounds in the nasal cavity.
3. Nasal cavity abnormalities that prevents catheter insertion.
4. A concomitant condition that could cause excessive nose bleeding or ongoing treatment with anticoagulant medication (except Aspirin and Clopidogrel).
5. A known allergy to polyurethane (polyurethane is used in the catheter balloon).
6. Systemic diseases with manifestations in the nose.
7. Previous treatment with radiation therapy to the nasal area.
8. Nasal surgery performed within the last six months.
9. Concurrent condition or risk of non-compliance that, in the investigator's opinion, may affect the interpretation of performance or safety data or which otherwise contraindicates participation in a clinical investigation;
10. Pregnant and lactating women;
11. Participation in a clinical investigation within 3 months of enrolment or planned participation at any time during this clinical investigation;
12. Previous participation in this study;
13. Employees of the study site or the sponsor directly involved with the conduct of the study, or immediate family members of any such individuals.

Only at baseline visit (day 0) If subject missed >4 days of eDiary entry, subject will be withdrawn.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of intranasal kinetic oscillation stimulation using the Chordate System S220 on monthly headache days with moderate to severe intensity after approx 6 weeks of treatment. | Baseline to 6 weeks
  Change in proportion of days with headache with moderate to severe intensity compared to the four week period starting the day after the third treatment Headache days are collected in electronic diary (eDiary)

SECONDARY OUTCOMES:
To evaluate the efficacy of treatment with KOS on monthly migraine days (regardless of intensity) Description: Migraine days are collected in an eDiary. | Baseline to 12 month
  Migraine days is collected in an eDiary.
To evaluate the incidence and severity of adverse events (AEs) and adverse device effects (ADEs) following treatment with the Chordate System S220. | Baseline to 12 month
  All adverse events (AEs) and adverse device effects (ADEs) incidence and severity following treatment with KOS
Number of patients who are responders | Baseline to 12 month
  Responders are classified as responder (less migraine/headache days) or non-responder (same or worsening of migraine/headache days).
  A responder is a patient who has decrease of headache/migraine days whilst a non responder had no or the same number of headache/migraine days
Number of patients who decrease use of abortive medication | Baseline to 12 month
  Intake of abortive medications are registered in eDiary and will be calculated on patient level
Mean change in Headache Impact Test (HIT-6) | Baseline to 12 month
  HIT-6 consist of 6 questions HIT-6 with scores from 6 to 13 where 13 is worst case per question so lower score is better outcome than high scores.
Mean change in Subject global severity | Baseline to 12 month
  Patient Global severity is a scale with four (4) scores, where normal (0) is the lowest and show no problems whilst severe (3) is the worst score 0. Normal
  1. Mild
  2. Moderate
  3. Severe

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Goadsby, Prof,MD,PhD, Principal Investigator — Wellcome Foundation Building, Denmark Hill Campus King's College London
Locations (12):
- Germany (4):
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden UniversitätsSchmerzCentrum, Dresden
  - Universitätsklinikum Essen (AöR) Klinik für Neurologie Kopfschmerz- und Schwindelambulanz, Essen
  - Kopfschmerzzentrum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Tübingen Klinik für Neurologie, Tübingen
- Shaare Zedek Medical Center, Neurology Clinics,, Jerusalem, Israel
- Italy (4):
  - IRCCS Istituto Auxologico Italiano U.O. Neurologia - Centro Cefalee, Milan
  - Centro Regionale Diagnosi e Cura delle Cefalee IRCCS National Neurological Institute "C. Mondino" Foundation, Pavia
  - Policlinico Universitario Campus Bio-Medico di Roma UOC Neurologia, Roma
  - IRCCS San Raffaele Pisana Dipartimento di Scienze Neurologiche Motorie e Sensoriali Unità per la Cura e la Ricerca su Cefalee e Dolore, Roma
- United Kingdom (3):
  - Department of Neurology, Institute of Neurological Sciences, Queen Elizabeth University Hospital, Glasgow
  - Hull Royal Infirmary, Hull University Teaching Hospital NHS Trust, Hull
  - St. George's University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Due to uncertainties in EU data protection legislation individual de-identified participant data are not shared. The main uncertainty is the concept of what "de-identified" means. It appears not to mean that the data set of a person is simply separated from the person's name. What additional operations have to be done appears to depend on technological capabilities to re-identify the persons associated with the data set. A common perception is that the technological capabilities for re-identification are permanently increasing. This could have the effect that public data sets that are regarded as de-identified now might become re-identifiable data sets in the future. Once this happens, the sponsor is no longer able to make the publication of the data sets un-happen. This could result in punishment by EU data protection authorities. The sponsor wants to avoid this.